CLINICAL TRIAL: NCT03142347
Title: Remote Endarterectomy vs Remote Endarterectomy Supplement DCB Balloon Angioplasty in Patients With the Femoral Artery Occlusive Disease (TASCII D)
Brief Title: Remote Endarterectomy vs Remote Endarterectomy + Drug Coated Balloon (DCB) Angioplasty in Patients With the Femoral Artery Occlusive Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-RICP-469
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Femoral Artery Occlusion
Keywords: remote endarterectomy; DCB balloon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote endarterectomy (Active Comparator): Open endarterectomy of the common, deep, initial of superficial femoral artery was performed. Delamination factory complex into the lumen of the loop. After that, the translational and rotational motions loops under fluoroscopic guidance, continuing detachment of plaque in the antegrade direction to the distal end of plaque. Plastic arteriotomy wounds performed patches of xenopericardium. Control patency of the arterial lumen is performed intraoperatively by X-ray angiography.
  Interventions: Procedure: Remote endarterectomy
- Remote endarterectomy + DCB balloon (Experimental): Open endarterectomy of the common, deep, initial of superficial femoral artery was performed. Delamination factory complex into the lumen of the loop. After that, the translational and rotational motions loops under fluoroscopic guidance, continuing detachment of plaque in the antegrade direction to the distal end of plaque. Plastic arteriotomy wounds performed patches of xenopericardium. And balloon angioplasty of superficial femoral artery with DCB balloon is perform. Control patency of the arterial lumen is performed intraoperatively by X-ray angiography.
  Interventions: Procedure: Remote endarterectomy + DCB balloon

INTERVENTIONS:
Procedure: Remote endarterectomy — Performed open endarterectomy of the common, deep, initial of superficial femoral artery. Proximal plaque exfoliate as far as possible in the superficial femoral artery. After that, the translational and rotational motions loops under fluoroscopic guidance, continuing detachment of plaque in the antegrade direction to the distal end of plaque. Plastic of arteriotomy wounds performed patches of xenopericardium. Control patency of the arterial vessel is performed intraoperatively by X-ray angiography. When rendering residual stenosis or intimal dissection, limiting blood flow, complemented by endovascular intervention plasticity.
  Arms: Remote endarterectomy
Procedure: Remote endarterectomy + DCB balloon — Performed open endarterectomy of the common, deep, initial of superficial femoral artery. Proximal plaque exfoliate as far as possible in the superficial femoral artery. After that, the translational and rotational motions loops under fluoroscopic guidance, continuing detachment of plaque in the antegrade direction to the distal end of plaque. Plastic of arteriotomy wounds performed patches of xenopericardium. And balloon angioplasty of superficial femoral artery with DCB balloon is perform. Control patency of the arterial vessel is performed intraoperatively by X-ray angiography. When rendering residual stenosis or intimal dissection, limiting blood flow, complemented by endovascular intervention plasticity.
  Arms: Remote endarterectomy + DCB balloon

SUMMARY:
Comparison effectiveness two methods revascularization of the superficial femoral artery: remote endarterectomy vs. remote endarterectomy supplemented DCB angioplasty in patients with steno-occlusive lesion of the femoro-popliteal segment of TASCII D

DETAILED DESCRIPTION:
Given that more and more devices appear to deliver cytotoxic drugs into the depth of atherosclerotic plaque, it is interesting to study the effect of these drugs when applied directly after plaque removal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with occlusive lesions of C and D type femoral artery and with chronic lower limb ischemia (II-IV degree by Fontaine, 4-6 degree by Rutherford)
* Patients who consented to participate in this study.

Exclusion Criteria:

* Chronic heart failure of III-IV functional class by New York Heart Association (NYHA) classification.
* Decompensated chronic "pulmonary" heart
* Severe hepatic or renal failure (bilirubin> 35 mmol / l, glomerular filtration rate <60 mL / min);
* Polyvalent drug allergy
* Cancer in the terminal stage with a life expectancy less than 6 months;
* Acute ischemic
* Expressed aortic calcification tolerant to remote endarterectomy
* Patient refusal to participate or continue to participate in the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
the change of lumen in target vessel | Baseline, 3 days after the operation, 6 month, 12 month, 2 years
  stenosis or occlusions

SECONDARY OUTCOMES:
Vessel wall thickness | 3 days after the operation, 6 month, 12 month, 2 years
  mm
Number of participants with limb salvage | 3 days after the operation, 6 month, 12 month, 2 years
Number of participants with complications in long-term period after the operation. | 3 days after the operation, 6 month, 12 month, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Karpenko, Study Director — cientific-Research Institute of Circulation Pathology named after Academician E. Meshalkin
Locations (1):
- Federal State Institution Academician E.N.Meshalkin Novosibirsk State Research Institute Of Circulation Pathology Rusmedtechnology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided